CLINICAL TRIAL: NCT01628120
Title: A Phase 3, Open-label, Multicenter, Long-term Safety Study Of Subcutaneous Epoetin Hospira In Patients With Chronic Renal Failure Requiring Hemodialysis And Receiving Epoetin Maintenance Treatment
Brief Title: A Phase 3, Long-Term Safety Study of Subcutaneous Epoetin Hospira in Patients With Chronic Renal Failure Requiring Hemodialysis and Receiving Epoetin Maintenance Treatment. AiME -Anemia Management With Epoetin
Acronym: AiME - 04
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPOE-11-04; C3461005 (Other: Alias Study Number)
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Results first posted 2018-07-19 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-02

CONDITIONS: Chronic Renal Failure Requiring Hemodialysis
Keywords: Chronic renal failure; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epoetin Hospira (Experimental): Epoetin Hospira will be administered by SC bolus injection 1 to 3 times per week per each patient's dosing schedule. Other ESAs (except for long-acting) may be used as rescue therapy.
  Interventions: Biological: Epoetin Hospira

INTERVENTIONS:
Biological: Epoetin Hospira — Subcutaneous(SC) injection
  Other Names: ESA; Erythropoetin Stimulation Agents

SUMMARY:
To determine the long term safety in treatment-emergent adverse events (TEAEs) of SC administration of Epoetin Hospira for maintenance of target hemoglobin (Hgb) levels in patients treated for anemia associated with chronic renal failure and on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to provide written Informed Consent after the risks and benefits of the study have been explained prior to any study related activities.
2. Patient previously completed the core study Maintenance Period up to and including Week 16 study assessments per protocol and is willing to continue open-label Epoetin Hospira for up to 48 weeks.
3. If female, patient must be postmenopausal for at least 1 year prior to enrollment, surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or practicing at least 1 of the following methods of birth control:

   * hormonal contraceptives (oral, parenteral, or transdermal) for at least 3 months prior to enrollment
   * intrauterine device
   * double-barrier method (condoms, contraceptive sponge, diaphragm, or vaginal ring with spermicidal jellies or cream)

   If hormonal contraceptives are used, the specific contraceptive must have been used for at least 3 months prior to enrollment. If the patient is currently using a hormonal contraceptive, she should also use a barrier method during this study and for at least 30 days following the administration of the patient's last open-label dose.
4. Adequate methods of contraception to prevent pregnancy are to be maintained throughout the course of the study in both male and female study subjects.

Exclusion Criteria:

1. Patient had a serious or severe adverse event in the core study that, in the opinion of the Investigator, was probably or definitely related to epoetin use and precluded safe use of epoetin.
2. Any of the following that developed during the core study and prior to enrollment:

   * Myocardial infarction
   * Stroke (cerebrovascular accident)/cerebrovascular insult (minor stroke) or transient ischemic attack/intracerebral bleeding/cerebral infarction
   * Severe/unstable angina
   * Coronary angioplasty, bypass surgery, or peripheral artery bypass graft
   * Decompensated congestive heart failure (New York Heart Association [NYHA] class IV)
   * Pulmonary embolism
   * Deep vein thrombosis or other thromboembolic event
   * Received live or attenuated vaccination (except flu vaccination)
3. A patient with any active, uncontrolled systemic, inflammatory, or malignant disease that developed during the core study and in the Investigator's opinion may be significant to exclude participation in the study, including but not limited to demyelinating diseases such as multiple sclerosis, microbial, viral, or fungal infection or mental disease.
4. Any newly developed significant drug sensitivity or a significant allergic reaction to any drug, as well as known hypersensitivity or idiosyncratic reaction to epoetin (or its excipients, including albumin) or any other related drugs that in the judgment of the Investigator is exclusionary for study participation.
5. A female patient who is pregnant, lactating, or planning a pregnancy during the study.
6. History of drug abuse or alcohol abuse during the core study prior to enrollment as determined by the Investigator.
7. Current participation or participation in a drug or other investigational research study within 30 days prior to enrollment (except the core study or any observational studies with prior written approval from Hospira).
8. May not be able to comply with the requirements of this clinical study, communicate effectively with study personnel, or is considered by the Investigator, for any reason, to be an unsuitable candidate for the study.
9. Evidence of human immunodeficiency virus (HIV) or hepatitis B surface antigen (HBsAg).
10. A patient who, in the Investigator's opinion, has any clinically significant abnormal laboratory results that may impact patient safety.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2012-05-31 (Actual); Primary Completion 2015-02-13 (Actual); Study Completion 2015-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (115):
- United States (115):
  - Azusa Dialysis Center, Azusa, California
  - Azusa, California
  - Pegasus Dialysis, Bakersfield, California
  - National Institute of Clinical Research, Bakersfield, California
  - Bakersfield, California
  - Bellflower Dialysis Center, Bellflower, California
  - Granada Hills, California
  - Lakewood Dialysis Center, Lakewood, California
  - Westcoast Dialysis, Long Beach, California
  - Long Beach Dialysis, Long Beach, California
  - Novo Research, Long Beach, California
  - Long Beach, California
  - Academic Medical Research Institute, Los Angeles, California
  - East LA Dialysis Center, Los Angeles, California
  - Los Angeles, California
  - Modesto Kidney Center, Modesto, California
  - Novo Research, Inc. d/b/a Foundation Research, Modesto, California
  - Parkway Kidney Center, Modesto, California
  - Modesto, California
  - US Renal Care of Northridge, Northridge, California
  - Northridge, California
  - Norwalk Dialysis Center, Norwalk, California
  - Oakdale Kidney Center, Oakdale, California
  - US Renal Care of Panorama City, Panorama City, California
  - Mohammad Ismail MD, Inc., Paramount, California
  - Paramount Dialysis Center, Paramount, California
  - Paramount, California
  - Canyon Country Dialysis Center, Santa Clarita, California
  - California Kidney Medical Group, Simi Valley, California
  - US Renal Care of Van Nuys, Van Nuys, California
  - intercommunity Dialysis Center, Whittier, California
  - American Institute of Research, Whittier, California
  - Whittier Kidney Dialysis Center, Whittier, California
  - Whittier, California
  - Kidney Center of Arvada, Arvada, Colorado
  - Western Nephrology and Metabolic Bone Disease, PC, Arvada, Colorado
  - Arvada, Colorado
  - Kidney Center of westminster, LLC, Westminster, Colorado
  - Western Nephrology and Metabolic Bone Disease, PC, Westminster, Colorado
  - Westminster, Colorado
  - Pines Clinical Research, Inc., Pembroke Pines, Florida
  - Pembroke Pines, Florida
  - Nephrology Centers of America - Augusta (NCA-A), Augusta, Georgia
  - Augusta, Georgia
  - Nephrology Centers of America (NCA) South Augusta, Augusta, Georgia
  - Kidney Care Associates, LLC, Augusta, Georgia
  - Grovetown Dialysis Center, Grovetown, Georgia
  - East Macon Dialysis, Macon, Georgia
  - Renal Physicians of Georgia, PC, Macon, Georgia
  - Macon, Georgia
  - Perry Dialysis Center, Perry, Georgia
  - Waynesboro Dialysis Center, Waynesboro, Georgia
  - Fresenius Medical Care Midtown #8498, Wichita, Kansas
  - Kansas Nephrology Research Institute, LLC, Wichita, Kansas
  - Wichita, Kansas
  - FMC Northside, Lafayette, Louisiana
  - Research Nurse Specialists ,LLC, Lafayette, Louisiana
  - Lafayette, Louisiana
  - FMC Opelousas, Opelousas, Louisiana
  - Fresenius Medical Care- Kalamazoo East, Kalamazoo, Michigan
  - Fresenius Medical Care - Kalamazoo, Kalamazoo, Michigan
  - Nephrology Center DBA Paragon Health PC, Kalamazoo, Michigan
  - Kalamazoo, Michigan
  - Fresenius Medical Care - Oshtermo, Kalamazoo, Michigan
  - Fresenius Medical Care- Gull Road, Kalamazoo, Michigan
  - Belton, Missouri
  - Dialysis Clinics, Inc. - Belton, Belton, Missouri
  - FMC Metro North Dialysis, Florissant, Missouri
  - FMC Normandy Dialysis, Normandy, Missouri
  - FMC St. Louis Regional Dialysis, Saint Ann, Missouri
  - Metro Hypertension and Kidney Center, St Louis, Missouri
  - St Louis, Missouri
  - Dialysis Clinic Incorporated, North Brunswick, New Jersey
  - North Brunswick, New Jersey
  - Kennedy Dialysis Center, Sewell, New Jersey
  - Kennedy Dialysis Center, Voorhees Township, New Jersey
  - Voorhees Township, New Jersey
  - College Point, New York
  - Flushing, New York
  - Trude Weishaupt Memorial Dialysis Center, Fresh Meadows, New York
  - Wake Dialysis Clinic, Raleigh, North Carolina
  - Wake Nephrology Associates, PA, Raleigh, North Carolina
  - Raleigh, North Carolina
  - DCI McMillan, Cincinnati, Ohio
  - Cincinnati, Ohio
  - Innovative Dialysis of Toledo, Toledo, Ohio
  - Toledo Hospital, Promedica Health System, Toledo, Ohio
  - Toledo, Ohio
  - Alexis Dialysis Center, Toledo, Ohio
  - Wildwood Dialysis Center, Toledo, Ohio
  - meadville Dialysis, Meadville, Pennsylvania
  - The Center for Hypertension and Nephrology Care, Meadville, Pennsylvania
  - Fresenius Medical Care, Knoxville, Tennessee
  - Cedar Bluff Dialysis, Knoxville, Tennessee
  - Knoxville Kidney Center, PLLC, Knoxville, Tennessee
  - Knoxville, Tennessee
  - Fresenius Medical Care-Austin North Dialysis, Austin, Texas
  - Research Management Inc., Austin, Texas
  - Research Management, Inc., Austin, Texas
  - Austin, Texas
  - Fresenius Medical Care - Cedar Park, Cedar Park, Texas
  - Grand Prairie Dialysis Center, Grand Prairie, Texas
  - Grand Prairie, Texas
  - Mission Bend Dialysis, Houston, Texas
  - Southwest Houston Research, Ltd., Houston, Texas
  - Houston, Texas
  - SNG Dialysis Center of Lufkin, Lufkin, Texas
  - Lufkin, Texas
  - San Antonio Kidney Disease Center Physicians Group, P.L.L.C., San Antonio, Texas
  - Las Palmas Davita Dialysis Center, San Antonio, Texas
  - San Antonio, Texas
  - ARA Mechanicsville Dialysis, Mechanicsville, Virginia
  - Nephrology Specialists, P.C., Mechanicsville, Virginia
  - Mechanicsville, Virginia
  - ARA South Laburnum Dialysis, Richmond, Virginia

REFERENCES:
- [Derived] Wish JB, Rocha MG, Martin NE, Reyes CRD, Fishbane S, Smith MT, Nassar G. Long-term Safety of Epoetin Alfa-epbx for the Treatment of Anemia in ESKD: Pooled Analyses of Randomized and Open-label Studies. Kidney Med. 2019 Aug 28;1(5):271-280. doi: 10.1016/j.xkme.2019.06.009. eCollection 2019 Sep-Oct. PMID 32734207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with chronic renal failure were receiving Epoetin maintenance therapy in study EPOE-10-13 (NCT01473420) prior to enrollment and treatment in the current study.
Groups:
- Epoetin Hospira: Participants were enrolled to receive Epoetin Hospira subcutaneous injection 1 to 3 times every week over a period of 48 weeks. Dose was adjusted to maintain the hemoglobin (Hb) level from 9 to 11 gram per deciliter (g/dL).
Period: Overall Study
Arm/Group | Epoetin Hospira
Started | 173
Treated | 170
Completed | 129
Not Completed | 44
Not completed — Withdrawal by Subject | 7
Not completed — Adverse Event | 12
Not completed — Lost to Follow-up | 1
Not completed — Not met Inclusion/Exclusion Criteria | 2
Not completed — Non-compliant with Study Procedures | 1
Not completed — Not Treated | 3
Not completed — Sponsor Decision | 5
Not completed — Switched Dialysis Method | 2
Not completed — Missed Study Drug More than 2 Weeks | 3
Not completed — Moved or Relocated | 5
Not completed — Kidney Transplant | 2
Not completed — Use of Standard of Care | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all enrolled participants who received at least 1 dose of Epoetin Hospira.
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.63 (12.903)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 75

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs): Week 1
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment emergent are events that emerged during the treatment period and were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Up through 7 days after first dose of study drug (Week 1)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of Epoetin Hospira. Here, "number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 167
Percentage of participants | 17.4

2. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs): Over Week 1 to 12
Description: as for outcome 1
Time Frame: Week 1 up to Week 12
Population: Safety analysis set included all enrolled participants who received at least 1 dose of Epoetin Hospira.
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 170
Percentage of participants | 67.1

3. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs): Over Week 13 to 24
Description: as for outcome 1
Time Frame: Week 13 up to Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 157
Percentage of participants | 60.5

4. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs): Over Week 25 to 36
Description: as for outcome 1
Time Frame: Week 25 up to Week 36
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 145
Percentage of participants | 57.9

5. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs): Over Week 37 to 48
Description: as for outcome 1
Time Frame: Week 37 up to Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 134
Percentage of participants | 48.5

6. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (AEs): Over Week 1 to 48
Description: as for outcome 1
Time Frame: Week 1 up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of Epoetin Hospira.
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 170
Percentage of participants | 87.6

7. Secondary Outcome: Mean Weekly Dosage of Epoetin Hospira: Over Week 1 to 48
Time Frame: Week 1 up to Week 48
Population: Full analysis set (FAS) included all enrolled participants and had at least 1 dose of Epoetin Hospira and had at least 1 Hb value.
Measure: Mean (Standard Deviation); unit: Unit per kilogram per week (U/kg/week)
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 169
Unit per kilogram per week (U/kg/week) | 83.74 (93.983)

8. Secondary Outcome: Mean Weekly Dosage of Epoetin Hospira for Interval of 12 Weeks
Time Frame: Week 1 up to Week 12; Week 13 up to Week 24; Week 25 up to Week 36; Week 37 up to Week 48
Population: FAS included all enrolled participants and had at least 1 dose of Epoetin Hospira and had at least 1 Hb value. Here, 'n' signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: U/kg/week
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 169
U/kg/week
  Week 1 to Week 12: number analyzed (Participants) | 167
  Week 1 to Week 12 | 80.49 (86.310)
  Week 13 to Week 24: number analyzed (Participants) | 154
  Week 13 to Week 24 | 83.14 (94.060)
  Week 25 to Week 36: number analyzed (Participants) | 142
  Week 25 to Week 36 | 85.98 (98.414)
  Week 37 to Week 48: number analyzed (Participants) | 131
  Week 37 to Week 48 | 88.86 (120.284)

9. Secondary Outcome: Mean Hemoglobin Levels: Over Week 1 to 48
Time Frame: Week 1 up to Week 48
Population: FAS included all enrolled participants and had at least 1 dose of Epoetin Hospira and had at least 1 Hb value.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 169
g/dL | 10.24 (0.553)

10. Secondary Outcome: Mean Hemoglobin Levels for Interval of 12 Weeks
Time Frame: Week 1 up to Week 12; Week 13 up to Week 24; Week 25 up to Week 36; Week 37 up to Week 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 169
g/dL
  Week 1 to Week 12 | 10.16 (0.735)
  Week 13 to Week 24: number analyzed (Participants) | 156
  Week 13 to Week 24 | 10.28 (0.636)
  Week 25 to Week 36: number analyzed (Participants) | 145
  Week 25 to Week 36 | 10.30 (0.717)
  Week 37 to Week 48: number analyzed (Participants) | 134
  Week 37 to Week 48 | 10.25 (0.791)

11. Secondary Outcome: Mean Hematocrit Levels: Over Week 1 to 48
Description: Hematocrit is defined as the percentage of red blood cells in the blood.
Time Frame: Week 1 up to Week 48
Population: FAS included all enrolled participants and had at least 1 dose of Epoetin Hospira and had at least 1 Hb value.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 169
Percentage of red blood cells | 32.22 (2.091)

12. Secondary Outcome: Mean Hematocrit Levels for Interval of 12 Weeks
Description: Hematocrit is defined as the percentage of red blood cells in the blood.
Time Frame: Week 1 up to Week 12; Week 13 up to Week 24; Week 25 up to Week 36; Week 37 up to Week 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 169
Percentage of red blood cells
  Week 1 to Week 12 | 31.90 (2.516)
  Week 13 to Week 24: number analyzed (Participants) | 156
  Week 13 to Week 24 | 32.32 (2.358)
  Week 25 to Week 36: number analyzed (Participants) | 145
  Week 25 to Week 36 | 32.40 (2.657)
  Week 37 to Week 48: number analyzed (Participants) | 134
  Week 37 to Week 48 | 32.31 (2.851)

13. Secondary Outcome: Percentage of Participants With Hemoglobin Level Outside Target Range
Description: Percentage of participants with hemoglobin level outside the target range of 9.0 to 11.0 g/dL were reported.
Time Frame: Week 1 up to Week 48
Population: FAS included all enrolled participants and had at least 1 dose of Epoetin Hospira and had at least 1 Hb value.
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 169
Percentage of participants | 86.4

14. Secondary Outcome: Percentage of Participants Who Received Blood Transfusions
Time Frame: Week 1 up to Week 48
Population: FAS included all enrolled participants and had at least 1 dose of Epoetin Hospira and had at least 1 Hb value.
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 169
Percentage of participants | 8.3

15. Other Pre Specified Outcome: Percentage of Participants With Hemoglobin Level Less Than (<) 8.0 Gram Per Deciliter (g/dL)
Time Frame: Week 1 up to Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 169
Percentage of participants | 13.0

16. Other Pre Specified Outcome: Percentage of Participants With Hemoglobin Level Greater Than (>) 12.0 Gram Per Deciliter (g/dL)
Time Frame: Week 1 up to Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 169
Percentage of participants | 20.7

17. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Hemoglobin (Hb) Levels
Description: Participants with clinically significant change from baseline in hemoglobin levels were upon investigator's discretion.
Time Frame: Baseline up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of Epoetin Hospira.
Measure: Number; unit: Participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 170
Participants | 0

18. Other Pre Specified Outcome: Number of Participants Who Received Concomitant Medication
Time Frame: Week 1 up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of Epoetin Hospira.
Measure: Number; unit: Participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 170
Participants | 170

19. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Tests
Description: Laboratory tests included: Hematology (hematocrit, hemoglobin, red blood cells count, reticulocytes, white blood cells count, neutrophils, bands, lymphocytes, monocytes, basophils, eosinophils, platelets, mean corpuscular volume); Coagulation panel (prothrombin time, international normalized ratio, activated partial thromboplastin time); Chemistry (blood urine nitrogen, creatinine, total bilirubin, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, sodium, potassium, magnesium, calcium, gamma-glutyl transpeptidase, phosphorus, uric acid, total protein, glucose, albumin, C-reactive protein); iron status (plasma ferritin, transferrin saturation). Participants with clinically significant change from baseline in laboratory tests were based on investigator's discretion.
Time Frame: Baseline up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of Epoetin Hospira.
Measure: Number; unit: Participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 170
Participants | 0

20. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in 12-Lead Electrocardiogram (ECG)
Description: ECG parameters included: PR interval, QRS complex, QT interval and QTC interval. Participants with clinically significant change from baseline in 12-lead ECGs were based on investigator's discretion.
Time Frame: Baseline up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of Epoetin Hospira.
Measure: Number; unit: Participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 170
Participants | 0

21. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examinations
Description: Physical examination included examination of the skin, eyes, ears, throat, neck, and cardiac, respiratory, gastrointestinal and musculoskeletal systems. The examination assessed the participants for any clinically significant changes in physical status, as determined by the investigator.
Time Frame: Baseline up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of Epoetin Hospira.
Measure: Number; unit: Participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 170
Participants | 0

22. Other Pre Specified Outcome: Percentage of Participants With Anti-Recombinant Human Erythropoietin (rhEPO) Antibodies
Description: Percentage of participants with at least 1 positive anti-rhEPO antibodies were reported. Radioimmunoprecipitation assay method was used to determine the presence of anti-rhEPO antibodies.
Time Frame: Baseline, Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of Epoetin Hospira. Here, "n" signifies those participants who were evaluable at specified time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Epoetin Hospira
Number analyzed (Participants) | 170
Percentage of participants
  Baseline | 0.6
  Week 48: number analyzed (Participants) | 144
  Week 48 | 0.7

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study. Safety population.
Arm/Group | Epoetin Hospira
Serious Adverse Events (participants affected / at risk) | 59/170
Other Adverse Events (participants affected / at risk) | 127/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Epoetin Hospira (N=170)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Bundle branch block left (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 3
Cardiac failure congestive (Cardiac disorders) | 6
Cardio-respiratory arrest (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Mitral valve stenosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Nodal rhythm (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Optic neuropathy (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Diabetic gastroparesis (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 2
Rectal fissure (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Appendicitis perforated (Infections and infestations) | 1
Arteriovenous graft site infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Enterococcal bacteraemia (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 5
Respiratory tract infection (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Staphylococcal sepsis (Infections and infestations) | 3
Sepsis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 2
Hip fracture (Injury, poisoning and procedural complications) | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 3
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Calciphylaxis (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/75 — This is a gender specific event.
Cerebral haemorrhage (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Hospira (N=170)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 27
Nausea (Gastrointestinal disorders) | 27
Headache (Nervous system disorders) | 25
Diarrhoea (Gastrointestinal disorders) | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 18
Dizziness (Nervous system disorders) | 17
Hypotension (Vascular disorders) | 17
Upper respiratory tract infection (Infections and infestations) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Fall (Injury, poisoning and procedural complications) | 13
Anaemia (Blood and lymphatic system disorders) | 11
Vascular graft complication (Injury, poisoning and procedural complications) | 11
Anxiety (Psychiatric disorders) | 10
Nasopharyngitis (Infections and infestations) | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 9
Oedema peripheral (General disorders) | 9
Pain (General disorders) | 9
Pyrexia (General disorders) | 9
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single centre publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.